CLINICAL TRIAL: NCT03497793
Title: A Feasibility Study of the SNUBY®, a Skin-to-skin Garment, in the Preterm Infant
Acronym: Preterm SNUBY®
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Contractual issues have halted study set up
Sponsor: University Hospitals of Derby and Burton NHS Foundation Trust (Other)
Collaborators: University of Birmingham (Other); University of Nottingham (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: DHRD/2017/097
Record Dates: First submitted 2018-03-16; First posted 2018-04-13 (Actual); Last update posted 2021-02-01 (Actual); Status verified 2021-01

CONDITIONS: Premature Birth; Breast Feeding
MeSH Terms: conditions — Premature Birth; Breast Feeding

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Skin-to-skin care with SNUBY (Experimental): Mothers providing skin-to-skin care with the use of SNUBY
  Interventions: Other: SNUBY

INTERVENTIONS:
Other: SNUBY — Following written informed consent, mother will be issued with an appropriate sized SNUBY® for her use only. The infant will be placed in skin-to-skin in SNUBY®, infant chest to mother's chest whilst the mother is seated on a reclining chair, allowing the infant to be further stabilised by gravity. Monitor wires, IV lines and/or ventilation tube will be secured using the ties on the SNUBY®. The infant's temperature, pulse and SaO2 will be recorded prior to skin-to-skin, repeated as required for the infant's clinical condition or at 30min intervals for the duration of skin-to-skin. Maternal and infant behaviour will be recorded, including spontaneous breastfeeding. The time taken to put the infant into skin-to-skin care, time in skin-to-skin care and time to return to cot will be recorded.

SUMMARY:
Skin-to-skin care (placing the nappy-clad baby on the mother's bare chest and draping both in a blanket) is known to benefit both baby and mother. Benefits to the baby include warmth, reduced crying, and stabilisation of heart rate, breathing and blood sugar, and promotion of breastfeeding while simultaneously reduces mother's anxiety, improves bonding, and increases breastmilk production. Although these benefits are even more pronounced for preterm, studies show most preterm babies do not receive adequate skin-to-skin care due to fears such as dislodging intravenous lines, ventilation tubes, monitor wires and concerns about safety and privacy. Measures are therefore required to increase maternal confidence and awareness and facilitate skin-to-skin care for preterm infants.

SNUBY® (SNUggle baBY) is a purpose-built garment for facilitation of skin-to-skin care in preterm infants. It is made of comfortable, breathable bamboo fabric with an attractive appearance such that it can be worn as a normal garment.

In addition, it has distinctive features that allow the baby to be placed in a specially designed pouch, in direct contact with the mother's skin, with supports for lines and tubes that may be attached to the baby. Although many garments are commercially available for mothers to carry babies, no such specially designed garment has ever been tested scientifically and none are specifically designed for preterm babies. In this observational study, the investigators will initially test the feasibility of using the SNUBY® in preterm infants by inviting five mothers-preterm infant pairs, with mother's written informed consent, to use the garment under direct supervision. Following this, the investigators will analyse the safety and acceptability of using it on a larger scale to facilitate skin-to-skin care in preterm babies. The investigators will gather information on the staff and mothers' knowledge of skin-to-skin care and their experience of using SNUBY®.

DETAILED DESCRIPTION:
Skin-to-skin contact is used as part of a package of Kangaroo Mother Care across the world. This has been demonstrated to reduce neonatal morbidity, mortality, and inpatient stays for low birth weight and preterm infants (Charpak and Ruiz 2016).

This study examines the effect a facilitating garment, the Snuby® has on neonatal health outcomes associated with skin-to-skin contact, such as neonatal thermoregulation, breastfeeding status, and self-reported mother-infant bonding. It uses a mixed methods approach to address quantitative and qualitative outcomes including participant's perspectives, and measurable health markers.

ELIGIBILITY:
Inclusion Criteria:

* Preterm (born at < 37 weeks gestation) infants
* Admitted to the Neonatal Intensive Care Unit
* Well enough to receive skin-to-skin care
* Mothers who agree to participate AND Mothers of eligible preterm infants

Exclusion Criteria:

*Any infant or mother considered unsuitable for skin-to-skin care for medical reasons (as decided by the attending Consultant Neonatologist).

Ages: 0 Days to 4 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Gender Based: Yes — Adult participants will be mothers - this is because the garment is desinged for women. In the future, modified garment will be desinged for use by fathers.
  Infants of both gender will be included in the study.
Enrollment: 0 (Actual)
Dates: Start 2021-12 (Estimated); Primary Completion 2021-12 (Estimated); Study Completion 2021-12 (Estimated)

PRIMARY OUTCOMES:
Infant's body temperature 30 minutes after starting skin-to-skin care with the SNUBY® | Following 30 minutes of skin-to-skin contact.
  Axillary temperature of the infant taken 30 min after starting skin-to-skin care
Infant's body temperature 30 minutes after completing skin-to-skin care with the SNUBY® | Following 30 minutes of skin-to-skin contact.
  Axillary temperature taken 30 minutes after completing skin-to-skin care
Number of episodes of desaturations (oxygen saturation levels below the cut off for infant's gestational age and postnatal age) and/or bradycardia (heart rate <100 beats per minute) | Following 30 minutes of skin-to-skin contact.
  discreet events of desaturations or bradycardia

SECONDARY OUTCOMES:
Mother's acceptability of the SNUBY® | Six weeks post birth.
  assessed by a five point Likert scale/visual analogue scale
Mother's comfort level while using SNUBY® | Six weeks post birth.
  assessed by a five point Likert scale/visual analogue scale
Neonatal staff's acceptability of the SNUBY® | 12 months post birth of the first participating mother-infant dyad.
  assessed by a five point Likert scale/visual analogue scale
Neonatal staff's ease of facilitating skin-to-skin care with SNUBY® | 12 months post birth of the first participating mother-infant dyad.
  assessed by a five point Likert scale/visual analogue scale

CONTACTS AND LOCATIONS:
Overall Officials: Shalini Ojha, Principal Investigator — Royal Derby Hosptial

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] 1. WHO. Preterm birth. Secondary Preterm birth 2016. http://www.who.int/mediacentre/factsheets/fs363/en/. 2. ONS. Birth Charactersitics. Secondary Birth Charactersitics 2016. https://www.ons.gov.uk/peoplepopulationandcommunity/birthsdeathsandmarriages/livebirths/datasets/birthcharacteristicsinenglandandwales. 3. Conde-Agudelo A, Diaz-Rossello JL. Kangaroo mother care to reduce morbidity and mortality in low birthweight infants. Cochrane Database Syst Rev 2016(8):CD002771. 4. Engmann C, Wall S, Darmstadt G, et al. Consensus on kangaroo mother care acceleration. Lancet 2013;382(9907):e26-7. 5. Seidman G, Unnikrishnan S, Kenny E, et al. Barriers and Enablers of Kangaroo Mother Care Practice: A Systematic Review. Plos One 2015;10(5).